CLINICAL TRIAL: NCT05977985
Title: The Effects of Rotator Interval Hydro-dissection in Primary Adhesive Capsulitis. A Two-arm Double-blind Randomised Controlled Trial
Brief Title: The Effects of Rotator Interval Hydro-dissection in Primary Adhesive Capsulitis.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023630-12612
Record Dates: First submitted 2023-07-19; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Adhesive Capsulitis of Shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dextrose 5% (Experimental): Rotator interval hydro-dissection with dextrose 5% solution
  Interventions: Drug: Rotator interval hydro-dissection with dextrose 5%
- Corticosteroid (Active Comparator): Rotator interval hydro-dissection with corticosteroid solution
  Interventions: Drug: Rotator interval hydro-dissection with corticosteroid solution

INTERVENTIONS:
Drug: Rotator interval hydro-dissection with dextrose 5% — Single injection of 20ml dextrose 5% into the rotator interval around the long head biceps tendon under ultrasound guidance using a 11-14 Hz frequency linear probe
  Arms: Dextrose 5%
Drug: Rotator interval hydro-dissection with corticosteroid solution — Single injection of 20ml corticosteroid solution (1 ml triamcinolone 40 mg/ml + 19 ml saline 0.9%) into the rotator interval around the long head biceps tendon under ultrasound guidance using a 11-14 Hz frequency linear probe
  Arms: Corticosteroid

SUMMARY:
Adhesive capsulitis (AC) is a significant cause of chronic shoulder pain and disability. Non-surgical option consisting of intraarticular corticosteroid (IA CS) injection with structured physiotherapy (PT) is the current standard of care. More recent randomized controlled trials have found that rotator interval (RI) hydro-dissection approach leads to better improvement in pain as compared to IA approach. Despite being non-inferior to surgical management, long-term outcome studies of patients treated with IA CS injection and PT have shown that patients only achieve satisfactory outcomes in 72.3% of patients after a mean symptom duration of 41.8 months. Furthermore, CS injections are associated with significant systemic and local adverse effects such as Cushing syndrome, osteopenia/ osteoporosis, infection, and hyperglycemia. In recent years, dextrose injection has emerged as an effective alternative to CS-based injections to treat chronic painful musculoskeletal conditions such as chronic low back pain, peripheral nerve entrapment and lateral epicondylitis.

The investigators aim to study the effects of RI hydro-dissection with dextrose 5% (D5%) on pain relief, shoulder ROM and shoulder function in patients with primary AC.

ELIGIBILITY:
Inclusion Criteria:

* patients with primary adhesive capsulitis
* aged 35 to 65 years of age
* duration of symptoms in between 3 to 18 months
* limitation in flexion, abduction, and external rotation greater than 30 degrees compared to normal
* limitation in internal rotation with hand to back shoulder test below L4

Exclusion Criteria:

* diagnosis of connective tissue disease or inflammatory arthritis
* history of surgery to the affected shoulder
* history of shoulder dislocation/ fracture
* neurological weakness of the affected upper limb
* ultrasound findings of rotator cuff or LHBT tendinopathy
* plain radiographs showing significant glenohumeral joint osteoarthritis (Kallgren-Lawrence grade 3 or 4)
* other sources of chronic pain
* bilateral adhesive capsulitis
* history of pain intervention to the shoulder joint in the past 3 months
* allergic reaction to local anesthetic agent

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Shoulder pain | 1 week, 4 weeks and 12 weeks post injection
  Shoulder pain based on Shoulder Pain and Disability Index (SPADI) pain scale. The SPADI pain scale ranges from 0 to 50, with higher score indicating greater level of pain.

SECONDARY OUTCOMES:
Shoulder range of motion | 4 weeks and 12 weeks post injection
  Shoulder range of motion in flexion, abduction, external rotation, internal rotation
Shoulder function | 4 weeks and 12 weeks post injection
  Shoulder function based on Shoulder Pain and Disability Index (SPADI) disability scale. The SPADI disability scale ranges from 0 to 80, with higher score indicating greater level of disability.

OTHER OUTCOMES:
Adverse events | from time to injection up till 1 week post injection
  Adverse events during or after injection